CLINICAL TRIAL: NCT03915015
Title: VAPORHCS/OHSU J: Safety of Clinically Indicated Magnetic Resonance Imaging in Patients With Permanent Pacemakers (PPM) and Implanted Cardioverter Defibrillators (ICDs)
Brief Title: VAPORHCS/OHSU J: MRI and Devices
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Charles Henrikson, MD, Professor of Medicine, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 8423
Record Dates: First submitted 2019-03-13; First posted 2019-04-16 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: MRI

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- the study (Other): Patients with a PPM or ICD getting a clinically indicated MRI
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — MRI

SUMMARY:
This is a database study of clinically indicated MRIs on patients with permanent pacemakers and implantable cardioverter defibrillators.

DETAILED DESCRIPTION:
1. Abstract

   Ferromagnetic Implants such as PPM's and ICD's are traditionally accepted as contraindications to MRI due to safety concerns. The hypothesis is that these procedures can be safely performed when appropriate safety precautions and vetting practices are implemented.

   This is a cohort study. 1000 patients with a clinical need for MRI will be included in the study at OHSU. The type of device and leads will be ascertained and a safety protocol will be strictly adhered to.
2. Background

   It has been estimated that 50-75% of patients with implanted devices (pacemakers and ICDs) will develop an indication for magnetic resonance imaging (MRI) examination. Thus, there are approximately 200,000 patients annually denied MRI scans because of the presence of PPMs and ICDs in the United States. The current standard of care is not to perform these scans, and instead to utilize other (inferior) imaging, and make clinical decisions without the benefit of MRI imaging. This is the current standard of care of OHSU, where only pacemaker patients who are not pacemaker dependent can undergo MRI scans, per radiology policy. However, this leads to gaps in care for some patients who would clearly benefit from an MRI scan. In some centers, it has been shown that when proper precautions are taken, MRIs can be safely performed on patients with PPMs and ICDs. The published experience from Johns Hopkins reports over 500 scans performed without any adverse outcomes.(1) There are also several smaller studies documenting the safe experience with MRI scanning in device patients (reviewed in (1), table 4)

   The main concerns which have led to restrictions on MRIs in patients with cardiac rhythm devices are the following:(2)
   1. Force and torque-ferromagnetic devices in a magnetic field are subject to static and gradient magnetic field induced force and torque. However, the maximum force that a modern PPM or ICD generator would be subject to is 100g, far under what would be needed to dislodge a device.
   2. Current induction-the gradient magnetic fields in the MRI scanner could induce current in conductors in the field. However, the maximum observed current in vitro has been less than 0.5mA, far less than what is required to capture myocardium.
   3. Heating-Leads and other metallic devices can act as antennae, and may heat in the magnetic field, however, no heating greater than 0.5deg C were observed in vitro.
   4. Inappropriate pacing/shock/inhibition of pacing-Pacemakers and ICDs have the possibility of receiving electromagnetic interference from the MRI and having this lead to inappropriate pacing, inhibition of pacing, ICD shocks, reprogramming, or loss of function.

   While all of the concerns are real and have been reported in earlier generation devices, with proper patient selection and monitoring during the scan, MRIs can be performed safely on most device patients. Johns Hopkins has an experience of over 500 scans without any adverse events.(1) The proposed protocol here follows exactly the Hopkins protocol, and, indeed, the OHSU data will be combined with the Hopkins data for future publications.

   To review the most recent Johns Hopkins publication:(1) 555 MRI studies in 438 device (PPM and ICD) patients were reported. All MRI scans were clinically indicated, and a device clinician, familiar with device interrogation and programming, was physically present for the entire duration of the scan. All patients were continuously monitored via telemetry and pulse oximetry during the MRI. For pacemaker patients, if they are pacemaker dependent they were reprogrammed to a non-sensing mode for the scan. If they were not pacemaker dependent, they were left in their usual mode. For ICD patients, if they were not pacemaker dependent, they were left in their usual mode. However, pacemaker dependent ICD patients were not scanned, as ICDs generally do not have a non-sensing pacing mode. Therapy for tachycardia was disabled in all ICDs for the scan.

   There were three clinical events during scans, all were "power on resets", which means that the device resets to "out of the box" original factory settings. One of these patients had an ICD, felt tugging in his chest during the scan, and the scan was not completed. The other two power on resets were in PPM patients, in whom the scan was completed. Neither were pacemaker dependent, and neither noticed anything abnormal during the scan. All three patients had normally functioning devices following the scan, and at followup.

   In the overall patient population in the Hopkins study, no single patient had a malfunction of a device immediately following the scan. There was a slight change in the electrical parameters of the leads, on average, but this did not result in the need for any intervention on any patient.
3. Objectives

   The primary objective of this study is to develop a protocol, consistent with DHHS/CMS guidelines and requirements to further document safety in clinically indicated MR imaging in patients with implanted cardioverter defibrillators (ICD's) and pacemakers.
4. Study Procedures

   MRI's will be conducted on patients who require a clinically indicated MRI only. All studies will be done in the 1.5 Tesla MRI unit. ECG monitoring pads will be placed on the patients for the duration of the study. An external defibrillator and ACLS drugs will be on hand. Heart rate, blood pressure, O2 saturation will also be monitored non-invasively throughout the study. All devices will undergo a complete interrogation prior to imaging. Parameters such as atrial and ventricular pacing thresholds, R and P wave amplitudes, lead impedance, and battery status will be measured and recorded. PPMs will be programmed to an asynchronous mode if dependent and to an inhibited mode in patients without pacemaker dependence.

   The pacemaker function of ICD's in pacemaker independent patients will be programmed to ventricular inhibited (VVI) mode at 50 bpm. Pacemaker dependent patients with ICDs will be excluded.

   In addition, there is a theoretical concern that patients who have capped or abandoned leads in their chest may be at risk for heating. While there is little or no objective data to support this concern, given this theoretical concern, patients in this category will only be admitted to the study if the referring physician deems the MRI critical and after the PI has carefully considered the risk/benefit ration for each patient who falls in to this category.

   Similarly, there historically has also been a concern that newly implanted leads (<4 weeks) are at risk for lead to dislodgement d/t possible torque from the MRI environment. This too is only a theoretical concern and there is little or no scientific evidence to support this claim. Nevertheless, patients with newly implanted pacemaker/ICD leads will be considered by the PI for protocol inclusion only if the referring physician deems the MRI to be critical and after considering the risk/benefit to each individual patient.

   After the appropriate MRI protocol for each MRI patient's unique condition has been completed, the device will be re-programmed to its original settings and completely interrogated to detect any changes in device performance.

   The duration of the study extends to the post procedure interrogation at 1-6 weeks post MRI. IF the PPM or ICD reveals any malfunction post imaging (not seen yet), the patient will be followed by the electrophysiology service and appropriate follow-up management will be arranged.
5. Study Statistics

   1. Primary outcome variable. Patient safety and device malfunction during or after MRI
   2. Secondary outcome variables. None
   3. Statistical plan including sample size justification and interim data analysis. We hope to enroll 1000 patients over 4 years to further evaluate safety.
   4. Early stopping rules. N/A
6. Risks

   1. Medical risks, listing all procedures, their major and minor risks and expected frequency.

      There are no studies showing any health hazards associated with magnetic field exposure. PPM and ICD implants subjected to the strong electromagnetic field of MR imaging are thought to be susceptible to movement and torque. Other traditional concerns include malfunction due to demagnetization or magnetic activation leading to inappropriate pacing and shocks and artificial sensing of electromagnetic interference from MRI leading to inappropriate inhibition and/or activation of antitachycardia therapy, device malfunction and induced arrhythmias, as detailed in the background section above. Heating of the device and surrounding tissues leading to fibrosis and increased capture thresholds have also been a theoretical concern. However, recent work has revealed the safety of PPM's and certain ICD's in the MR environment given appropriate precautions(1, 3, 4).
   2. Steps taken to minimize the risks. Appropriate measures discussed in the protocol section will be taken to minimize risks associated with device exposure to MRI. Consistent with standard MRI policy, patients in the first trimester of pregnancy and patients with history of allergic reactions to gadolinium will undergo imaging without any contrast media.
   3. Plan for reporting unanticipated problems or study deviations. Patient data will be monitored on a per patient basis. Pre-vs. post MRI device testing data will be compared and any significant differences immediately reported to the IRB.
7. Benefits a. Description of the probable benefits for the participant and for society. The patient will benefit from a standardized protocol to minimize the risk of an MR scan deemed necessary for his/her care which would otherwise be denied or performed without any organized framework. Society will benefit because of the increasing number of implanted devices and expanding use of MRI.

8 Costs

a. Detail costs of study procedure(s) or drug (s) or substance(s) to participants and identify who will pay for them.

The patient and his/her insurance will be responsible for the cost of the clinically indicated MRI.

ELIGIBILITY:
Inclusion Criteria:

- Patients with an absolute clinical need for MR imaging and PPM (year 1996 model or later) or ICD's (year 2000 or later)

Exclusion Criteria:

* Patients with pacemaker models before 1996 and ICD models before year 2000.
* Pacemaker dependent patients with ICD.
* Patients who weighing less than 80 lbs.
* Patients who complete the MRI standard screening form and are deemed inappropriate for MRI for any reason
* Pregnant patients will be excluded in their first trimester and will not get gadolinium at any time during their pregnancy
* Patient with abandoned/capped leads or leads implanted <4 weeks unless the procedure is deemed critical by the referring physician and approved by the PI

Ages: 9 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2012-07-19 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
MRI Safety during MRI scan in patients with PPMs/ICDs. | During MRI scan.
  Percent of patients successfully completing MRI scan without complication per interrogation of their device and clinical assessment.
MRI Safety following MRI scan in patients with PPMs/ICDs. | 1-6 week follow up in device clinic
  Percent of patients successfully following up after MRI scan without complication per interrogation of their device and clinical assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Henrikson, MD, Principal Investigator — Oregon Health and Science University
Locations (2):
- United States (2):
  - Oregon Health and Scince University, Portland, Oregon
  - Portland Veterans Administration Medical Center, Portland, Oregon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yadava M, Nugent M, Krebsbach A, Minnier J, Jessel P, Henrikson CA. Magnetic resonance imaging in patients with cardiac implantable electronic devices: a single-center prospective study. J Interv Card Electrophysiol. 2017 Oct;50(1):95-104. doi: 10.1007/s10840-017-0262-6. Epub 2017 Jul 22. PMID 28733766
- [Background] Nazarian S, Hansford R, Roguin A, Goldsher D, Zviman MM, Lardo AC, Caffo BS, Frick KD, Kraut MA, Kamel IR, Calkins H, Berger RD, Bluemke DA, Halperin HR. A prospective evaluation of a protocol for magnetic resonance imaging of patients with implanted cardiac devices. Ann Intern Med. 2011 Oct 4;155(7):415-24. doi: 10.7326/0003-4819-155-7-201110040-00004. PMID 21969340